CLINICAL TRIAL: NCT05781204
Title: "Perceived Stigma and Social Support: Relationship and Influence on Mental Health and Quality of Life in HIV+ Patients"
Brief Title: Stigma, Social Support and Quality of Life
Acronym: 4826
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: SPESS
Record Dates: First submitted 2023-01-30; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Each participant completed an anonymous 62-item online survey.

SUMMARY:
The primary goal of this observational study is to investigate the relationship between perceived stigma and social support in HIV+ patients. The secondary objective is to measure mental health indicators (depression, anxiety, and stress) and quality of life to assess whether they are affected by the relationship between perceived stigma and social support.

The main questions it aims to answer are:

* Measuring perceived stigma and social support to understand the health status and behaviour of people living with HIV.
* Monitor the mental state of people living with HIV in order to be able to implement, there where necessary, a psychological support strategy in order to promote proper adherence to treatment and care services.

Participants will fill out an online cross-sectional survey. The online questionnairesurvey will collect:

* sociodemographic and clinical data related to HIV infection,
* perceived stigma,
* social support,
* mental health,
* quality of life.

ELIGIBILITY:
Inclusion Criteria:

* HIV diagnosis.
* Being treated at the Infectious Diseases Outpatient Clinic of Policlinico Gemelli in Rome.
* Ongoing antiretroviral therapy.
* Age > 18 years.
* Native Italian speaker.
* Informed consent to participate in the study.

Exclusion Criteria:

* Absence of an HIV diagnosis.
* Not being treated at the Infectious Diseases Outpatient Clinic of Policlinico Gemelli in Rome.
* Absence of ongoing antiretroviral therapy.
* Age > 18 years.
* Not being a native Italian speaker.
* Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We expect the majority of the HIV patient population to be male, between the ages of 40 and 65 and with a high school diploma. We expect a virologically suppressed HIV population with good adherence to antiretroviral therapy. We expect a high level of perceived stigma and low quality of life and high symptoms of depression, anxiety and stress.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Perceived stigma in HIV+ patients | 1 year
  Perceived stigma in HIV+ patients will be assess through the following test: the 12-item short version of the HIV stigma scale. The test consists of four subscales: personalized stigma, concerns about disclosure of one's HIV status, concerns about the attitudes of others and negative self-image.

SECONDARY OUTCOMES:
Influence of social support on perceived stigma | 1 year
  HIV+ patients' perceived social support will be examined through the use of 6 statements (1. "If you are sick, you have someone to rely on physically for example as help with household chores or as company during doctor's visits"; 2. "You have someone who can look after your home if you are away"; 3. "If you wanted to go on a trip, you would have someone to share the experience with"; 4. "You have someone who accepts you with your strengths and faults"; 4. "You have someone who loves you and gives you affection"; 6. "If you have emotional difficulties, you have someone who listens to you and gives you support and advice").
Influence of mental health on perceived stigma | 1 year
  Mental health will be investigated using the Depression Anxiety Stress Scale (DASS) 21, a self-assessment instrument containing 21 useful items to investigate three constructs: depression, anxiety and stress. Each construct constitutes a specific subscale, consisting of 7 items. Each item corresponds to a statement, referring to the past week.
Influence of quality of life on perceived stigma | 1 year
  Quality of life will be investigated using the 12-item Short-Form Health Survey (SF-12). The SF-12 investigates quality of life with 12 items: 6 items are concerned with physical health (physical functioning, physical plane limitations, physical pain, general health) and 6 items are concerned with mental health (emotional plane limitations, fatigue or lack of energy, social functioning, emotional well-being).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No